CLINICAL TRIAL: NCT02415543
Title: A Prospective, Randomized, Controlled Trial of Comparing Single Incisional Laparoscopic Total Extraperitoneal(SIL-TEP) Inguinal Hernia Repair With Traditional Laparoscopic Total Extraperitoneal(TEP) Inguinal Hernia Repair in Day Surgery
Brief Title: SIL-TEP vs TEP for Inguinal Hernia Repair in Day Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TAO CHEN (Other)
Responsible Party: Sponsor-Investigator, TAO CHEN, attending doctor, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RenJi Hospital
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP A (Active Comparator): Group A will undergo SIL-TEP inguinal hernia repair with a single port LESS (12 to 15 mm paraumbilical)
  Interventions: Procedure: SIL-TEP Inguinal Hernia Repair
- GROUP B (Active Comparator): Group B will undergo laparoscopic TEP inguinal hernia repair with 3 ports (10 mm , and 2 ports of 5 mm )
  Interventions: Procedure: TEP Inguinal Hernia Repair

INTERVENTIONS:
Procedure: SIL-TEP Inguinal Hernia Repair — perform the laparoscopic total extraperitoneal inguinal hernia repair using a single incision
  Other Names: SIL-TEP repair
  Arms: GROUP A
Procedure: TEP Inguinal Hernia Repair — perform the multiport laparoscopic total extraperitoneal inguinal hernia repair
  Other Names: TEP repair
  Arms: GROUP B

SUMMARY:
This study aim to compare the efficacy and safety of Single incisional Laparoscopic Total Extraperitoneal(SIL-TEP) Inguinal Hernia Repair and traditional Laparoscopic Total Extraperitoneal(TEP) Inguinal Hernia Repair in day surgery. This study also aim to improve the surgical-related technical details and the device design.

In addition, this study also evaluate the operability of SIL-TEP in term of a day surgery item and try to provide the basis for SIL-TEP day surgery guildline, so as to promote the SIL-TEP technology in the investigators country.

DETAILED DESCRIPTION:
This is a prospective, randomized，controlled trail. It compared Single Incisional Laparoscopic Total Extraperitonea(SIL-TEP) with traditional Laparoscopic Total Extraperitoneal(TEP) Inguinal Hernia Repair in condition of day surgery.

Laparoscopic hernia repair technique including two tyes, TEP and TAPP, which were recognized as mordern minimally invasive technique. Laparoscopic hernia repair were recommended by the Association of Surgeons of Great Britain and Ireland (ASGBI) and European Hernia Society Guideline (EHS) as the first choice for primary inguinal hernia. Compared with TAPP, TEP was performed much more frequently for its advantages of avoiding abdominal visceral injury.

Traditional TEP hernia repair involves 3-port insertions: one incision of 2cm in para-umbilical region for the camera and two smaller incisions of 5mm each in the midline for the surgical instruments. Some surgeons think the second and third ports could led to bowel and bladder injury. Early literatures showed that bowel injuries and bladder injuries were observed in TAPP or TEP hernia repair.

Since 2009, Cugura JF and Filipovic-Cugura J led their teams for a preliminary exploration of SIL-TEP. Later, several cases were reported about this surgical technique globally. Since then, a number of retrospective studies about the comparation of SIL-TEP and traditional TEP were carried. Yang GP et al found that SIL-TEP had a longer operation time than traditional TEP, but in terms of postoperative complications and incision aesthetics. Tu Wenbin et al thought that SIL-TEP was effective and also had advantages in postoperative pain, postoperative complications and time in hospital. Several other reports also had similiar opnions.

However, randomized controlled trial related to this suject is quite limited. Our study aim to compare the efficacy and safety of SIL-TEP and traditional TEP surgery with a RCT design and also aim to improve the surgical-related technical details and the device design. Our study also evaluate the operability of SIL-TEP in term of a day surgery item and try to provide the basis for SIL-TEP day surgery guildline, so as to promote the SIL-TEP technology in our country.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of primary unilateral inguinal hernia and age between 18 and 70 ;
2. Good condition of family care and observation, understand and be willing to accept day surgery mode;
3. Willing to participate in this study and signed an informed consent.

Exclusion Criteria:

1. Diagnosed as femoral hernia, recurrent hernia, scrotal hernia, bilateral hernia and strangulated hernia;
2. Patients with severe chronic diseases or cardiopulmonary dysfunction;
3. American Society of Anesthesiologists (ASA) grade III and IV level;
4. Obese patients ( BMI> 30 );
5. Patients with a history of lower abdominal surgery;
6. prefer to a centain surgical approach.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
SIL-TEP Conversion to TEP / TAPP or open operation | during operation
  This refers to whether any SIL-TEP procedure needs to be converted to TEP/TAPP or open procedure. This is quite a normal process as a proportion of multiport procedures are converted to open procedures for safety reasons.

SECONDARY OUTCOMES:
Operating time | during operation
  This assess the time taken to perform the operation and is defined as time from initial skin incision to complete wound closure
interoperation complication | during operation
  Assessment of interoperation procedure of the incident of spermaduct、vessel and other organ damage
Pain score (Visual Analog Scale) at 12、24 hour and one week after surgery | 12、24hour and day 7 postoperation
  Assessment of post-operative pain according to the visual analog scale Pain score will be taken, and any painkiller consumption will be recorded
Length of hospital stay | 1 day postoperation
  This assess how long patients stay in hospital and whether it is a day surgery or they need to extend time stay in hospital
return to work or normal physical activities | 4 weeks postoperation
  Patients will be followed up and assesses how soon patients return to normal physical activities and work
Cosmetic scar score | 4 weeks
  Patients will be followed up and asked to assess satisfaction of their own scars 4 weeks postoperation
post-operative complications including urinary retention, wound infection, wound haematoma，seroma formation, chronic pain, testicular atrophy | 1 week, 4 weeks after postoperation
  Patients will be followed up and assessed at 1 week, 4 weeks after surgery to assess for any post-operative complications associated with hernia surgery as enumerated above
Recurrence of hernia | 4 weeks，3 mounths and 1 year postoperation
  Patients will be followed up and assessed at 4 weeks，3 mounths and one year after surgery to detect the presence of recurrence of hernia
hospitalization costs | 1 day postopetation
  Hospitalization costs will be assessed after operation at discharge form the hospital

CONTACTS AND LOCATIONS:
Overall Officials: JIAN WANG, MD, Study Chair — Director of Biliary and Pancreatic Surgery Department Renji Hospital, Shanghai Jiao Tong University, School of Medicine
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided